CLINICAL TRIAL: NCT04609397
Title: A Phase Ⅱ Study to Evaluate the Efficacy and Safety of Hemay005 in the Treatment of Behçet Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Hemay005 in the Treatment of Behçet Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study purpose has been achieved
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HM005BD2S01
Record Dates: First submitted 2020-10-19; First posted 2020-10-30 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Behçet Disease
Keywords: Behçet Disease
MeSH Terms: conditions — Behcet Syndrome | interventions — Hemay005; Cyclic Nucleotide Phosphodiesterases, Type 4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemay005 high dose group (Experimental): In Core-treatment period, subject will take Hemay005 60mg twice daily for 12 weeks, and in the following extend-treatment period, subject will take Hemay005 60mg twice daily for 12 weeks.
  Interventions: Drug: Hemay005
- Hemay005 lower dose group (Experimental): In Core-treatment period, subject will take Hemay005 45mg twice daily for 12 weeks, and in the following extend-treatment period, subject will take Hemay005 45mg twice daily for 12 weeks.
  Interventions: Drug: Hemay005
- Placebo (Placebo Comparator): In Core-treatment period, subject will take placebo for 12 weeks, and in the following extend-treatment period, subject will take Hemay005 60mg or hemay005 45mg twice daily according to pre-allocation at randomization visit for 12 weeks.
  Interventions: Drug: Hemay005; Other: Placebo

INTERVENTIONS:
Drug: Hemay005 — Hemay005 tables 60mg bid p.o;
  Other Names: Phosphodiesterase 4 (PDE4) inhibitors
  Arms: Hemay005 high dose group; Placebo
Drug: Hemay005 — Hemay005 tables 45mg bid p.o
  Other Names: Phosphodiesterase 4 (PDE4) inhibitors
  Arms: Hemay005 lower dose group; Placebo
Other: Placebo — placebo to Hemay005 tables bid p.o
  Arms: Placebo

SUMMARY:
This is a phase 2, multi-center, randomized, placebo-controlled, double-blind, parallel-group study with an equal randomization among the Hemay005 high dose, lower dose and placebo treatment groups. After subject randomization, each subject will enter an core-treatment Phase for 12 weeks following an extended-treatment phase for another 12weeks and a follow up phase for 4weeks.

DETAILED DESCRIPTION:
this study is a phase 2, multi-center, randomized, placebo-controlled, double-blind, parallel-group study to evaluate Hemay005 efficacy and safety of the treatment of patients with Behçet Disease(BD). Around 252 subjects will be randomized into this study.

The whole study will including 4 phases that a screening phase, core-treatment phase(12weeks), extended-treatment phase (12weeks) and follow-up phase(4 weeks).

Screening: All subjects will undergo a screening period of up to 6 weeks prior to baseline visit (visit 2, day of randomization, Day0).

Core treatment phase: eligible BD patients will randomly assigned to Hemay005 high-dose group, Hemay005 low-dose group, placebo (core treatment phase) + Hemay005 high-dose group (extended treatment phase), or placebo (core treatment phase) + Hemay005 low-dose group (extended treatment phase). During the core-treatment period, hemay005 will be administered twice daily for 12 weeks. The randomization was stratified to minimize the imbalance between treatment groups.

Extended treatment phase: Subjects in the high-dose and low-dose groups during the extended treatment period will still given the dose of core-treatment phase for 12 weeks. Subjects who received placebo during the core treatment will assigned to either a high-dose group or a low-dose group according the allocation at visit 2 until 12 weeks after. During this period, the subject and investigator are remain blind at this stage.

Follow up phase: Subjects in the study (also including those who withdraw from treatment for any reason) will have another follow up for 4 weeks after the end of the last administration.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understand and voluntarily sign an informed consent form prior to any study related assessments/procedures being conducted.
* 2.Male and female subjects 18~75(inclusive) years of age at the time of signing the informed consent form.
* 3.Diagnosed with Behçet's disease meeting the International Study Group (ISG) criteria (2013).
* 4.Subjects must have at least 2 oral ulcers at V1, and:

  1. at least 2 oral ulcers at V2 if V2 occurs at least 14 days after Visit 1, OR
  2. at least 3 oral ulcers at V2 if V2 occurs at least 0~42 days after Visit 1.
* 5. According to the site investigator judgement, subject is suitable to the systemic but not topical treatment of oral ulcer considering the severity and affected area of the disease OR the oral ulcer cannot be well controlled by topical treatment and have to take the systemic treatment.
* 6.All females of childbearing potential (FCBP) and male subjects who did not receive the vasectomy must take effective contraceptive measures.

Exclusion Criteria:

* 1.subject has the BD related major organ activity lesions requiring immunosuppressive therapy- pulmonary, vascular, gastrointestinal, and central nervous systems (eg, meningoencephalitis) manifestations, etc. However:

  1. Previous major organ involvement is allowed if it occurred at least one years prior to screening visit and is not active at time of enrollment.
  2. Subjects with BD-related arthritis and BD-skin manifestations are also allowed
* 2. Any clinically significant heart disease (e.g., but not limited to unstable ischemic heart disease, New York Heart Association(NYHA) class III / IV left ventricular failure, or myocardial infarction) or clinically significant 12 lead ECG abnormalities found during screening, which, according to the investigator's judgment, may put the patient at safety risk or may interfere with the investigator;
* 3. subjects who current receiving immunotherapy including:

  1. 7 days prior to Visit 2 (randomization) for colchicine.
  2. 10 days prior to Visit 2 (randomization) for azathioprine, mycophenolate mofetil, baricitinib or Tofacitinib.
  3. 4 weeks prior to visit 2(randomization) for cyclosporin, methotrexate, cyclophosphamide, thalidomide, and dapsone.
  4. At least 5 terminal half-lives for all biologics, including,within:

     1. Four weeks prior to visit 2(randomization) for etanercept.
     2. Eight weeks prior to visit 2(randomization) for infliximab.
     3. Ten weeks prior to visit 2(randomization) for adalimumab, golimumab, abatacept, and tocilizumab.
     4. Six months prior to visit 2(randomization) for secukinumab.
* 4.Having received intra-articular or parenteral corticosteroids within 6 weeks (42 days) prior to Visit 2.
* 5.Laboratory examination of V1 in screening period:

  1. Hemoglobin ≤ 85g / L;
  2. The white blood cell (WBC) count was less than 3.0 × 10^9 / L or more than 14 × 10^9 / L;
  3. Platelet < 100 × 10^9 / L;
  4. Serum creatinine > 1.5mg/dl (> 132.6 μ mol / L);
  5. Total bilirubin > 2.0 mg / dl (> 34.2 μ mol / L);
  6. The Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) were higher than 1.5 times of the upper limit of normal value.
* 6.subjects who received strong cytochrome P450 enzyme inducer within 4 weeks prior to visit2.
* 7.Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C and herpes zoster, histoplasmosis, coccidiomycosis, but excluding onychomycosis) , judged by investigator,may put the patient at safety risk.
* 8.Clinically significant abnormality on chest radiograph or CT,judged by investigator, may put the patient at safety risk.
* 9.History of transplantation and immunodeficiency disease, including those subject has a positive test for human immunodeficiency virus (HIV).
* 10.subject who use of any investigational products of clinical trials within 4 weeks or within 5 pharmacokinetic/pharmacodynamic half-lives prior to randomization, whichever is longer;
* 11.known to be allergic or allergic to the investigational products or ingredients;
* 12.History of alcohol or drug abuse, or a history of mental illness;
* 13.Subjects with severe, progressive, or uncontrolled disease, judged by the investigator, who maybe at risk if participate this study or those subjects whose participation may influence the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
to evaluate the efficacy of Hemay005 in the treatment of Behçet's disease. | week 12
  Area under the curve (AUC) for the number of oral ulcers from baseline through Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving an oral ulcer complete response | week 6
  Proportion of subjects achieving an oral ulcer complete response (oral ulcer-free) by Week 6 after dosing, and who remain oral ulcer free for at least 6 additional weeks during the Treatment Phase
Complete response rate for oral ulcers | day 3, day 7 and week12
  Complete response rate for oral ulcers at day 3, day 7 and Week 12
change of the pain evaluation of oral ulcers as measured by Visual analogue scale(VAS)(From 0-100, the higher score means the worse outcome) | week12
  Change from baseline in the pain of oral ulcers as measured by VAS at Week 12
change of the number of oral ulcers | week12
  Change from baseline in the number of oral ulcers at Week 12
Time to oral ulcer resolution | week12
  Time to oral ulcer resolution (complete response) that the first instance when a subject has a complete response during the core-Treatment Phase
Proportion of subjects achieving an oral ulcer complete response in the core-treatment phase | week12
  Proportion of subjects achieving an oral ulcer complete response (oral ulcer-free) and who remain oral ulcer free during the core-treatment Phase
Number of oral ulcers who has a reappearance during the core-treatment phase | week12
  Number of oral ulcers following loss of complete response that the first instance when a subject has a reappearance of oral ulcers following a complete response during the core-Treatment Phase
Time to oral ulcer reappearance during the core-treatment | week12
  Time to recurrence of oral ulcers following loss of complete response that the first instance when a subject has a reappearance of oral ulcers following a complete response during the core-Treatment Phase
change of the total score of Physician's Global Assessment(PGA) | week12
  change from baseline in the total score of the PGA of skin lesions of BD at week 12 in those subjects who had at baseline
change of BD Current Activity Form(BDCAF) | week12
  change from baseline in the total score of the BDCAF questionnaire at week 12
change of Multi-Dimensional Health Assessment Questionnaire (MDHAQ) | week12
  change from baseline in the total score of the MDHAQ questionnaire at week 12
change of short from health survey(SF-36) | week12
  change from baseline in the total score of the SF-36 questionnaire at week 12
Complete response rate for genital ulcers | week12
  Complete response rate for genital ulcers at Week 12 for subjects who had genital ulcers at Baseline
change of the pain evaluation of genital ulcers | week12
  Change from baseline in the pain of genital ulcers as measured by VAS at Week 12
Change of the Behçet's syndrome activity score(BSAS) score | week12
  Change from Baseline in BSAS score at Week 12
Maximum Plasma Concentration (Cmax) | week24
  the population pharmacokinetic (popPK) characteristics Cmax of Hemay005 in BD patients
Minimum Plasma Concentration (Cmin) | week24
  the population pharmacokinetic (popPK) characteristics Cmin of Hemay005 in BD patients
Time to peak (Tmax) | week24
  the population pharmacokinetic (popPK) characteristics Tmax of Hemay005 in BD patients
Elimination half-life (T1/2) | week24
  the population pharmacokinetic (popPK) characteristics T1/2 of Hemay005 in BD patients
Area under drug time curve (AUC) | week24
  the population pharmacokinetic (popPK) characteristics AUC of Hemay005 in BD patients
Clearance (Cl) | week24
  the population pharmacokinetic (popPK) characteristics Cl of Hemay005 in BD patients
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | week24
  the Incidence of Treatment-Emergent Adverse Events of Hemay005 in BD patients with different dosing group
the number of subjects who terminated hemay005 prematurely due to adverse events (AE) [Safety and Tolerability]) | week24
  the number of subjects who terminated hemay005 prematurely due to adverse events (AE) in BD patients with different dosing group

CONTACTS AND LOCATIONS:
Overall Officials: zhanguo Li, Doctor, Principal Investigator — Peking University People's Hospital
Locations (31):
- China (31):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui provincial hospital, Hefei, Anhui
  - Beijing hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-Sen Memorial Hospital,Sun Yat-Sen University, Guangzhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College of Inner Mongolia University of science and technology, Baotou, Inner Mongolia
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiu Jiang NO.1 people's Hospital, Jiujiang, Jiangxi
  - Jiangxi Pingxiang people's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - Linyi people's Hospital, Linyi, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital Of Tongji University Tang Jianping, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No